CLINICAL TRIAL: NCT02281253
Title: Evaluation of a Bakery Product Enriched With Fibre and L-carnitine on Cardiovascular Risk Parameters in Patients With Metabolic Syndrome: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Effects of a Bakery Product Enriched With Fibre and L-carnitine on Insulin Resistance in Patients With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Collaborators: AINIATechnology Center (Unknown)
Responsible Party: Principal Investigator, Antonio Hernandez Mijares, PhD, MD, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PAN-CAR-2010-01
Record Dates: First submitted 2014-10-28; First posted 2014-11-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Metabolic X Syndrome; Overweight; Dyslipidemias
Keywords: L-carnitine; fibre; bakery product; insulin resistance
MeSH Terms: conditions — Metabolic Syndrome; Overweight; Dyslipidemias; Insulin Resistance | interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- With metabolic syndrome (Experimental): Before dietary therapy was initiated, in order to stabilise dietary patterns prior to intervention, patients were submitted to a 4-weeks run-in period of a caloric restriction of 500 Kcal to their usual diet. After this adaptation period, two intervention groups were evaluated: a calorie-restricted diet plus bread-enriched product that received 15.08 g of dietary fibre (9.49 g of insoluble fibre and 5.59 g of soluble fibre) plus 2325 mg of L-carnitine/day in 130 g of bread (enriched group) and a calorie-restricted diet plus placebo bread group whose diet included 130 g/day of not-enriched bread (placebo group).
  Interventions: Dietary Supplement: dietary fibre plus L-carnitine bread; Dietary Supplement: Placebo bread
- Without metabolic syndrome (Experimental): Before dietary therapy was initiated, in order to stabilise dietary patterns prior to intervention, patients were submitted to a 4-weeks run-in period of a caloric restriction of 500 Kcal to their usual diet. After this adaptation period, two intervention groups were evaluated: a calorie-restricted diet plus bread-enriched product that received 15.08 g of dietary fibre (9.49 g of insoluble fibre and 5.59 g of soluble fibre) plus 2325 mg of L-carnitine/day in 130 g of bread (enriched group) and a calorie-restricted diet plus placebo bread group whose diet included 130 g/day of not-enriched bread (placebo group).
  Interventions: Dietary Supplement: dietary fibre plus L-carnitine bread; Dietary Supplement: Placebo bread

INTERVENTIONS:
Dietary Supplement: dietary fibre plus L-carnitine bread — The enriched bread consisted of a mix of wheat flour, vegetable flour, rye flour, wheat gluten, soy protein, soluble and insoluble dietary fibre, inulin, guar gum, L-carnitine salt, diacetyl tartaric, enzymes, ascorbic acid, water and yeast.
  Patients were recommended to consume the bread twice per day with main meals.
Dietary Supplement: Placebo bread — The placebo group received commercially available bread with a similar macronutrient composition and energy intake to that consumed by the enriched bread group but without L-carnitine and dietary fibre. Patients were recommended to consume the bread twice per day with main meals.

SUMMARY:
The aim of this study was to evaluate the efficacy of a bakery product enriched with dietary fibre and L-carnitine on glucose homeostasis and insulin sensitivity in overweight patients with or without metabolic syndrome.

DETAILED DESCRIPTION:
Conceivably, different biochemical changes in insulin-mediated signalling pathways may contribute to an impaired insulin-mediated glucose transport and metabolism that eventually results in insulin resistance and the clinical features of metabolic syndrome. According to this, both compounds -L-carnitine and dietary fiber- interacting by different mechanism of action could improve glucose homeostasis and insulin sensitivity. However, the health beneficial effects of the combination of both compounds are not shown and confirmation of the functionality of such products must be accomplished by conducting the appropriate studies intervention nutrition.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 35 Kg/m2

Exclusion Criteria:

* Pregnancy or lactation
* Kidney, liver and thyroid disease
* History of cardiovascular or chronic inflammatory disease
* Diabetes mellitus
* Lipid-lowering medication
* Triglyceride concentration > 400 mg/dl
* Consumption of other carnitine and/or fibre-enriched foods

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To assess changes in hydrocarbonated metabolism parameters before and after fibre+carnitine/placebo administration | baseline and 12 weeks
  Blood samples were collected in vacutainer serum separator tubes, after 12-hour overnight fasting, to analyze glucose, insulin and C-peptide concentration at baseline (after a four weeks run-in period of a healthy diet), and 12 weeks after fibre+carnitine/placebo administration.
  Glucose was determined using enzymatic techniques and insulin and C-peptide were measured by an enzymatic luminescence technique in an autoanalyzer. Insulin resistance was calculated by homeostasis model assessment (HOMA = (fasting insulin (μU/mL×) fasting glucose (mg/dl)/405).

SECONDARY OUTCOMES:
To evaluate changes in lipid parameters before and after fibre+carnitine/placebo administration | baseline and 12 weeks
  Blood samples were collected in vacutainer serum separator tubes, after 12-hour overnight fasting, to analyze lipid profile at baseline (after a four weeks run-in period of a healthy diet), and 12 weeks after fibre+carnitine/placebo administration. Total cholesterol and triglycerides were measured by means of enzymatic assays, and high-density lipoproteins (HDL) concentrations were recorded with an autoanalyzer using a direct method. Low-density lipoprotein (LDL) concentration was calculated using the method of Friedewald. Non-HDL concentration was obtained by calculating the difference between total cholesterol and HDL. LDL subfractions were separated by high-resolution polyacrylamide gel tubes. The LDL electrophoretic profile allows 2 patterns to be defined: pattern A or large and buoyant LDL, and pattern non-A or small and dense LDL.
To evaluate changes in a composite measure of inflammatory parameters before and after fibre+carnitine/placebo administration | baseline and 12 weeks
  Blood samples were collected in vacutainer serum separator tubes, after 12-hour overnight fasting, to analyze inflammatory markers at baseline (after a four weeks run-in period of a healthy diet), and 12 weeks after fibre+carnitine/placebo administration. Levels of high-sensitive C-reactive protein (hsCRP) and proinflammatory cytokines interleukin-6 (IL-6) and tumor necrosis factor-α (TNF-α) were analysed using a flow analyser system

OTHER OUTCOMES:
To assess adverse reactions after fibre+carnitine/placebo administration | 12 weeks
  Diarrhea, constipation, nausea, belching, flatulence, indigestion and bloating were evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hernández, Phd, MD, Principal Investigator — FISABIO - University Hospital Dr Peset

REFERENCES:
- [Background] Ringseis R, Keller J, Eder K. Role of carnitine in the regulation of glucose homeostasis and insulin sensitivity: evidence from in vivo and in vitro studies with carnitine supplementation and carnitine deficiency. Eur J Nutr. 2012 Feb;51(1):1-18. doi: 10.1007/s00394-011-0284-2. Epub 2011 Dec 2. PMID 22134503
- [Background] Malaguarnera M, Vacante M, Avitabile T, Malaguarnera M, Cammalleri L, Motta M. L-Carnitine supplementation reduces oxidized LDL cholesterol in patients with diabetes. Am J Clin Nutr. 2009 Jan;89(1):71-6. doi: 10.3945/ajcn.2008.26251. Epub 2008 Dec 3. PMID 19056606
- [Background] Sola R, Bruckert E, Valls RM, Narejos S, Luque X, Castro-Cabezas M, Domenech G, Torres F, Heras M, Farres X, Vaquer JV, Martinez JM, Almaraz MC, Anguera A. Soluble fibre (Plantago ovata husk) reduces plasma low-density lipoprotein (LDL) cholesterol, triglycerides, insulin, oxidised LDL and systolic blood pressure in hypercholesterolaemic patients: A randomised trial. Atherosclerosis. 2010 Aug;211(2):630-7. doi: 10.1016/j.atherosclerosis.2010.03.010. Epub 2010 Mar 17. PMID 20413122
- [Background] Robertson MD, Wright JW, Loizon E, Debard C, Vidal H, Shojaee-Moradie F, Russell-Jones D, Umpleby AM. Insulin-sensitizing effects on muscle and adipose tissue after dietary fiber intake in men and women with metabolic syndrome. J Clin Endocrinol Metab. 2012 Sep;97(9):3326-32. doi: 10.1210/jc.2012-1513. Epub 2012 Jun 28. PMID 22745235
- [Background] Gonzalez-Ortiz M, Hernandez-Gonzalez SO, Hernandez-Salazar E, Martinez-Abundis E. Effect of oral L-carnitine administration on insulin sensitivity and lipid profile in type 2 diabetes mellitus patients. Ann Nutr Metab. 2008;52(4):335-8. doi: 10.1159/000151488. Epub 2008 Aug 19. PMID 18714152